CLINICAL TRIAL: NCT02861859
Title: A Randomized Trial of Individualised Care Versus Standard Care for Breast Cancer Patients at High Risk for Chemotherapy Induced Nausea and Vomiting. The ILIAD Study
Brief Title: Individualised Versus Standard Care for Breast Cancer Patients at High-risk for Chemotherapy-induced Nausea and Vomiting The ILIAD Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTT 16-05
Record Dates: First submitted 2016-07-13; First posted 2016-08-10 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast Carcinoma; Breast Tumors; Chemotherapy; Antiemetic effects; Antiemetic drugs; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator): Eligible patients at high personal risk of CIVN will receive Standard of Care Regimen: Aprepitant (125 mg PO OD day 1, 80mg OD days 2-3), ondansetron (8mg PO, BID on Day 1 of each cycle), dexamethasone (12 mg IV x1 before chemotherapy and 4mg PO BID days 2-3) and olanzapine placebo (PO OD days 1-4).
  Eligible patients at low personal risk of CIVN will receive Standard of Care Regimen: Ondansetron (8mg PO, BID on Day 1 of each cycle,), dexamethasone (12 mg IV x1 before chemotherapy and 4mg PO BID days 2-3) and olanzapine placebo (PO OD days 1-4).
  Interventions: Drug: Olanzapine Placebo
- Olanzapine (Active Comparator): Eligible patients at high personal risk of CIVN will receive Standard of Care Regimen: Aprepitant (125 mg PO, OD day 1, 80mg OD days 2-3), ondansetron (8mg PO, BID on Day 1 of each cycle), dexamethasone (12 mg IV x1 before chemotherapy and 4mg PO BID days 2-3) and olanzapine (5 mg PO OD days 1-4).
  Eligible patients at low personal risk of CIVN will receive Standard of Care Regimen: Ondansetron (8mg PO, BID on Day 1 of each cycle), dexamethasone (12 mg IV x1 before chemotherapy and 4mg PO BID days 2-3) and olanzapine (5 mg PO OD days 1-4).
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5 mg (2 x 2.5 mg) PO OD (once a day) on days 1-4.
  Other Names: Mylan-Olanzapine
  Arms: Olanzapine
Drug: Olanzapine Placebo — Olanzapine Placebo 5 mg (2 x 2.5 mg) PO OD (once a day) on days 1-4.
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate whether adding olanzapine 5mg to standard antiemetic medication can significantly reduce chemotherapy-induced nausea and vomiting in breast cancer patients receiving emetogenic chemotherapy regimens such as anthracycline with cyclophosphamide-based chemotherapy and platinum-based chemotherapy.

To help clinicians prescribe antiemetic medications in a more patient-centered, evidence-based and cost-effective manner, we've developed the world's first validated risk-stratification tool for chemotherapy-induced nausea and vomiting (CINV) and because of this, it is now possible to perform a trial of personalized precision antiemetic therapy for breast cancer patients.

Despite widespread antiemetic use, chemotherapy-induced nausea and vomiting (CINV) remains among the most feared and expected side effects of chemotherapy for breast cancer. Inadequately controlled CINV can significantly reduce a patient's quality of life, impair functional activity, lead to chemotherapy dose delays and reductions, and even discontinuation of treatment. The merit of current antiemetic medications is based on their ability to control chemotherapy-induced vomiting, but not necessarily nausea, and nausea is the major issue for breast cancer patients.

With olanzapine demonstrating significant promise in preventing acute and delayed nausea, the investigators are proposing to evaluate guideline-recommended aprepitant-based triple regimen compared to the same regimen plus olanzapine (5 mg) for patients at high personal risk for CINV. For patients at low personal risk for CINV the investigators will also evaluate guideline-recommended double antiemetic regimen compared to the same regimen plus olanzapine (5 mg).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed invasive breast cancer (stage I-III) scheduled to receive neo/adjuvant anthracycline/cyclophosphamide or platinum-based chemotherapy
* ≥18 years
* Able to provide consent and complete all study-related diaries and questionnaires.

Exclusion Criteria:

* Received previous chemotherapy
* Symptoms of nausea or vomiting at baseline
* On chronic antiemetic therapy (e.g. metoclopramide); on daily long term oral steroids prior to chemotherapy
* Allergic or having a medical condition that makes the administration of olanzapine, aprepitant, 5-HT3 antagonists or dexamethasone contraindicated
* Uncontrolled diabetes
* Known/documented medical/psychiatric illness that would interfere with patients' ability to complete the diary and study-related questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-12; Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
High personal risk of Chemotherapy-induced nausea and vomiting | 3 years
  To assess whether the addition of olanzapine to the standard antiemetic regimens significantly reduces the incidence of nausea during the overall period, over repeated cycles of chemotherapy in patients at high personal risk for Chemotherapy-induced nausea and vomiting

SECONDARY OUTCOMES:
High personal risk overall total control of Chemotherapy-induced nausea and vomiting | 3 years
  To compare overall total control of Chemotherapy-induced nausea and vomiting (i.e. no nausea, no vomiting and no use of rescue medications) between the two study arms in the high risk cohort.
Improvement of patient Health Related Quality of Life by completing a patient diary and quality of life questionnaire in the high risk cohort | 3 years
  To assess whether adding olanzapine to a standard antiemetic regimen significantly improves patient Health Related Quality of Life in the high risk cohort
Safety of olanzapine with respect to sedation and extrapyramidal side effects in the high risk cohort | 3 years
  To assess the safety of adding olanzapine as a standard antiemetic regimen particularly with respect to sedation and extrapyramidal side effects in the high risk cohort

OTHER OUTCOMES:
Low personal risk of Chemotherapy-induced nausea and vomiting | 3 years
  To assess whether the addition of olanzapine to the standard antiemetic regimens significantly reduces the incidence of nausea in patients at personal low-risk for Chemotherapy-induced nausea and vomiting over repeated cycles of chemotherapy.
Low personal risk overall total control of Chemotherapy-induced nausea and vomiting | 3 years
  To compare overall total control of CINV (i.e. no nausea, no vomiting and no use of rescue medications) between the two study arms in the low risk cohort.
Improvement of patient Health Related Quality of Life by completing a patient diary and a quality of life questionnaire in the low risk cohort | 3 years
  To assess whether adding olanzapine to a standard antiemetic regimen significantly improves patient Health Related Quality of Life in the low risk cohort.
Safety of olanzapine with respect to sedation and extrapyramidal side effects in the low risk cohort | 3 years
  To assess the safety of adding olanzapine as a standard antiemetic regimen particularly with respect to sedation and extrapyramidal side effects in the low risk cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Research Institute Cance Center, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No